CLINICAL TRIAL: NCT00835302
Title: Development of a Clinical Prediction Rule to Identify Patients With Shoulder Pain Likely to Benefit From Cervicothoracic Manipulation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-0220; 1543340
Record Dates: First submitted 2009-02-02; First posted 2009-02-03 (Estimated); Last update posted 2013-01-30 (Estimated); Status verified 2009-02

CONDITIONS: Shoulder Pain
Keywords: Cervical; Thoracic; Manipulation; Mobilization; Clinical prediction rule; Shoulder pain.
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Manipulation + Exercise Group (Experimental): Cervicothoracic manipulation and ROM exercises
  Interventions: Procedure: Cervicothoracic manipulation

INTERVENTIONS:
Procedure: Cervicothoracic manipulation — Thrust and non-thrust manipulation to the cervical and thoracic spine
  Other Names: Mobilization

SUMMARY:
The investigators seek to develop a clinical prediction rule (CPR) to identify patients with a primary complaint of shoulder pain who are likely to benefit from manual therapy to the neck and upper back regions. Manual therapy will include mobilizations (therapist moves the joints in an oscillating fashion) and manipulations (therapist performs a high velocity low amplitude movement) The investigators hypothesize that a cluster of signs and symptoms from the subject history and physical examination will exist that maximize the accuracy of identifying patients with a primary complaint of shoulder pain likely to benefit from this manual therapy treatment based on a reference standard of patient-reported improvement.

The investigators also seek to investigate the psychometric properties (how good a test is), including test retest reliability of a modified version of the Fear Avoidance Beliefs Questionnaire (FABQ) and the shortened Tampa Scale for Kinesiophobia (TSK-11) in patients with shoulder pain. The investigators will also look at the convergent validity (determine if measures that should be related are in reality related) and discriminant validity (show that measures that should not be related are in reality not related) of the modified FABQ and the TSK-11 in patients with shoulder pain.

DETAILED DESCRIPTION:
The point prevalence of shoulder symptoms has been reported to range from 20-33% and the incidence of shoulder complaints in the general population is increasing. Furthermore, several authors have reported low rates of perceived recovery (patient reports of "being cured") for patients with a new episode of shoulder or neck pain.3-6 According to Bot et al, less than 25% of patients with a first episode of shoulder pain reported recovery after 3 months, and only 32% stated they had recovered (no longer had symptoms) after 1 year. Other studies have investigated the prognosis of shoulder pain in general practice. Croft et al reported recovery rates of only 21% after 6 months and 49% after 18 months. Van der Windt et al and Winters et al reported recovery rates of 51% and 59% after 12 to 18 months, respectively. Finally, Rekola et al reported that 25% of patients with shoulder or neck pain experienced at least one episode of recurrence within 12 months. These findings suggest that shoulder pain can be recurrent and frequently progresses to the chronic stage.

The Guide to Physical Therapist Practice describes 5 components of patient management; examination, evaluation, diagnosis, prognosis, interventions and outcomes. Information collected during the examination is evaluated in an attempt to improve decision making regarding the most appropriate treatment strategy for the individual patient. Contrary to the medical model which attempts to identify pathology to arrive at a diagnosis, the diagnostic process in physical therapy involves classifying or labeling patients based on functional limitations (restrictions in activities caused by a certain condition) and impairments (loss or abnormality in function such as decreased strength or motion) in an attempt to specifically direct treatment. Clinical decision making regarding treatment involves a certain degree of uncertainty as to which interventions will maximize individual patient outcomes. While the amount of quality evidence supporting physical therapy interventions is increasing, this uncertainty can make it difficult to decide on an appropriate treatment strategy. The American Physical Therapy Association has stated that identifying subgroups of patients who are likely to benefit from specific treatments is a research priority. (APTA) The Guide to Physical Therapist Practice indicates that interventions such as mobilization/manipulation are utilized by physical therapists to manage patients who have shoulder pain. There is growing evidence that impairments in the cervicothoracic spine may contribute to shoulder pain, and that patients with shoulder pain may benefit from manipulation in this region. Manipulation is defined as a manual therapy technique comprising a continuum of skilled passive movements, including small-amplitude/high velocity movements (thrust) and oscillations (non-thrust), that is targeted at joints and soft tissues.

While it is not likely that all patients who have with shoulder pain will benefit from manipulation (thrust and non-thrust) of the cervicothoracic spine, it is possible that a subgroup exists that will experience rapid and dramatic improvement with the use of these manual physical therapy techniques. It is our specific aim to develop a clinical prediction rule (CPR) to identify patients with a primary complaint of shoulder pain who are likely to benefit from cervicothoracic manipulation. The purpose of a CPR is to improve the clinician's accuracy in predicting a diagnosis or an expected outcome. For example, CPRs exist to improve the accuracy of diagnosing ankle fractures in individuals with acute injuries,predict the likelihood of death within four years for individuals with coronary disease, or determine when cervical radiographs are required for patients who have experienced neck trauma. The process of developing and testing a CPR has been described in detail elsewhere. Although CPRs can be developed to improve the accuracy of making a certain diagnosis, the focus of this project is to develop a CPR to predict a certain treatment outcome. The development of a CPR utilizes diagnostic properties of sensitivity, specificity, and positive and negative likelihood ratios, which are based on the individual patient. Thus their interpretation can be readily applied to an individual patient. Development of a CPR to accurately predict which patients with shoulder pain will likely experience a clinically meaningful improvement in pain and function with cervicothoracic spine manipulation before treatment would be immensely helpful for clinicians in the decision-making process. Thus the purpose of this project is to develop a CPR to identify patients with shoulder pain likely to benefit from cervicothoracic spine thrust and non-thrust manipulation.

ELIGIBILITY:
Inclusion Criteria:

* Primary complaint of shoulder pain (defined as pain between the neck and the elbow at rest or during movement of the upper arm, see diagram at right)
* Age between 18-65 years old
* Shoulder Pain and Disability Index (SPADI) score greater than 20 points (full description of this measure provided in self report measures section)

Exclusion criteria:

* Medical red flags noted in the patient's Medical Screening Questionnaire(i.e. tumor, fracture, metabolic diseases, RA, osteoporosis, weight loss, fever, prolonged history of steroid use, etc.)
* Acute fractures in the shoulder region.
* Acute severe trauma to the cervical (neck) or thoracic (upper back) regions in the last 6 weeks.
* Contraindications to manipulative therapy (for example osteoporosis of the cervicothoracic spine).
* Evidence of central nervous system involvement, to include hyperreflexia, sensory disturbances in the hand, intrinsic muscle wasting of the hands, unsteadiness during walking, nystagmus, loss of visual acuity, impaired sensation of the face, altered taste, the presence of pathological reflexes (i.e. positive Hoffman's and/or Babinski reflexes), etc.
* Diagnosis of cervical spinal stenosis or bilateral upper extremity symptoms
* Two or more positive neurologic signs consistent with nerve root compression, including any two of the following:

Muscle weakness involving a major muscle group of the upper extremity Diminished upper extremity muscle stretch reflex (biceps brachii, brachioradialis, or triceps brachii reflexes) Diminished or absent sensation to pinprick in any upper extremity dermatome

* Prior surgery to the neck or thoracic spine involving fusion or open reduction internal fixation.
* Insufficient English language skills to complete all questionnaires as they have only been validated in English.
* Inability to comply with treatment and follow-up schedule

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2006-10; Primary Completion 2008-12 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Global Rating of Change (GROC) | 7 days

SECONDARY OUTCOMES:
Shoulder Pain and Disability Index (SPADI) | 7 days
Numerical Pain Rating Scale | 7 days
Painfree Shoulder Range of Motion | 7 days

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - University of Colorado Denver, Aurora, Colorado
  - Wardenburg Health Center, Boulder, Colorado
  - Physiotherapy Associates, Greenwood Village, Colorado
  - Newton Wellesley Hospital, Newton, Massachusetts
  - Groves Physical Therapy, Saint Paul, Minnesota
  - Concord Hospital, Concord, New Hampshire

REFERENCES:
- [Derived] Mintken PE, Cleland JA, Whitman JM, George SZ. Psychometric properties of the Fear-Avoidance Beliefs Questionnaire and Tampa Scale of Kinesiophobia in patients with shoulder pain. Arch Phys Med Rehabil. 2010 Jul;91(7):1128-36. doi: 10.1016/j.apmr.2010.04.009. PMID 20599053
- [Derived] Mintken PE, Cleland JA, Carpenter KJ, Bieniek ML, Keirns M, Whitman JM. Some factors predict successful short-term outcomes in individuals with shoulder pain receiving cervicothoracic manipulation: a single-arm trial. Phys Ther. 2010 Jan;90(1):26-42. doi: 10.2522/ptj.20090095. Epub 2009 Dec 3. PMID 19959652